CLINICAL TRIAL: NCT02962687
Title: Video-Enhanced Care Management for Medically Complex Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PPO 15-425
Record Dates: First submitted 2016-10-25; First posted 2016-11-11 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Multimorbidity; Cognitive Impairments
Keywords: Veterans; Cognitive impairments; Nursing care management; Videoconferencing
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Videoconference care management (Experimental): 12-week nurse care management for medically complex Veterans with CI delivered via videoconferencing
  Interventions: Behavioral: Care management via videoconference
- Telephone care management (Active Comparator): 12-week nurse care management for medically complex Veterans with CI delivered via telephone calls
  Interventions: Behavioral: Care management via telephone calls

INTERVENTIONS:
Behavioral: Care management via videoconference — 12-week nurse care management for medically complex Veterans with CI delivered via videoconference
  Arms: Videoconference care management
Behavioral: Care management via telephone calls — 12-week nurse care management for medically complex Veterans with CI delivered via telephone calls
  Arms: Telephone care management

SUMMARY:
The purpose of this study is to examine the feasibility and acceptability of a 12-week care management program for medically complex Veterans with cognitive impairment, delivered via telephone or videoconferencing.

DETAILED DESCRIPTION:
BACKGROUND Older adults with complex care needs constitute a large and rapidly expanding group of Veterans receiving care within Veterans Health Administration (VHA). Medically complex older Veterans, who often have multiple chronic conditions (MCC) as well as interacting functional and psychosocial challenges, account for a disproportionate amount of health care resources. Importantly, these Veterans also experience a disproportionate amount of suffering; they have worse functional status, higher symptom burden, and spend more of their time in acute care settings such as the hospital and emergency department.

The investigators' experience and recent studies suggest that a substantial proportion of older medically complex Veterans have unrecognized cognitive impairment (CI), and this contributes to their disproportionate need for care and adverse outcomes. The Cumulative Complexity model posits that complexity results from accumulating and interacting clinical and social factors that each contribute to a patient's workload (e.g. making appointments and managing complicated medicine regimens) as well as impact a patient's capacity to perform everyday tasks including those related to health care. Imbalance between the two- i.e. workload that exceeds capacity-is a primary driver of disruptions in care and negative outcomes. Older patients with MCC, high health care utilization, and CI often find themselves in the perfect storm of complexity, simultaneously experiencing escalated workload demands in the setting of reduced capacity.

OBJECTIVES

The primary objectives of this pilot study are to:

Examine the feasibility and acceptability of a 12-week care management program for medically complex Veterans with CI, delivered via telephone or through video visits.

* Feasibility will be examined by calculating overall rates of eligibility and enrollment, as well as rates of attrition, adherence to nurse calls or video visits, and interview completion.
* Acceptability will be assessed using in-depth interviews with study participants (Veterans and Care Partners), primary care providers, and study staff.

Assess the usability and perceived value of video-enhanced care management, compared to telephone-based, among older Veterans with medical complexity and CI.

* Usability of the video-enhanced program will be examined using the System Usability Scale (SUS).
* Perceived value associated with each delivery method will be explored through questionnaires and in-depth interviews with study participants and study staff.

METHODS Veterans aged 65 or older with high medical complexity based on Care Assessment Need (CAN) score will be screened for CI using a reliable and valid instrument developed for use over the telephone. Veterans with CI, and a self-identified Care Partner, will participate in a nurse-led care management program designed to provide structured cognitively-appropriate information and support in two key areas: (1) care coordination (reduce workload) and (2) protecting cognitive health (build capacity). Evidence-based strategies to improve care coordination and promote cognitive health are enhanced by video visits that allow for improved communication between the nurse and Veteran/Care Partner, and facilitate expanded assessments of the Veteran and his/her home environment. Study measures will include the SUS, participant feedback, and measures of intervention effectiveness including health and physical function (PROMIS 29), physical activity levels (PASE), depression (PHQ-9), anxiety (GAD-7), and acute care days (hospital and ER).

ANTICIPATED IMPACT Results from this preliminary study will be used to inform the development of a randomized clinical trial to evaluate the impact of a 12-month video-enhanced care management program for medically complex older adults with CI. Given the large number of medically complex Veterans affected by unrecognized CI, it is essential that interventions targeting this population be scalable, and technology-enhanced interventions offer a way to expand the reach of new care models. Proactive recognition and management of medically complex patients is a high priority for VHA, and medically complex Veterans with CI constitute one such high risk group. The results of this study will be of high relevance to VHA, and outside VA, given the urgent need to develop innovative means of improving care for medically complex older adults.

ELIGIBILITY:
Inclusion Criteria:

* Receive primary care from a Durham Veterans Affairs Medical Center (VAMC) affiliated primary care clinic (1 visit within the previous 12 months)
* Age > or = 65
* CAN score > or = 90
* Valid telephone number in the medical record
* Identifies a friend or family member that we may contact for study participation as the Care Partner
* Telephone Instrument for Cognitive Status - modified (TICS-m) score 20-31

Exclusion Criteria:

* Cognitive impairment or dementia (identified via ICD diagnosis codes or Primary Care Provider note in previous 2 years)
* Enrolled in or have an active consult for a special population Patient Aligned Care Teams (PACT), e.g.:

  * GeriPACT
  * Home Based Primary Care
  * Mental Health
  * Post-Deployment, etc.
* Serious mental illness defined as diagnosis of psychosis of any type:

  * schizophrenia
  * bipolar disorder
  * psychiatric hospitalization in the previous year
  * or current high-risk suicide flag in their Computerized Patient Record System (CPRS) medical record
* Active substance abuse, documented in the medical record within the previous year
* Eligible for hospice, palliative care, or prognosis of less than 6 months to live
* Lacks decision-making capacity, documented in the medical record
* Referred to institutional care or residing in nursing home
* Unable to communicate on the telephone, or no telephone access for duration of study
* Currently hospitalized or incapacitated
* Enrolled in a study that prohibits participation in another study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan N. Hastings, MD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be available upon request. Prior to distribution, a local privacy officer and study statistician will certify that the dataset contains no protected health information (PHI). Data will be provided to requestor in electronic format.
  Sufficient data and descriptors will be made available to duplicate statistical analysis and confirm conclusions in publication.
  No data or statistical code that could lead to re-identification of individuals will be released.
  Data will be stored & maintained in an approved, secured location as described in the VA Research Data Inventory Form.
  The study statistician will create de-identified, publication-specific datasets that includes all variables presented in the study publication.
  Data will only be released per appropriate authorizations or agreements. Written agreements will specify that recipients are prohibited from taking steps to re-identify any individual whose data are included in the dataset.

RESULTS

PARTICIPANT FLOW:
Groups:
- Videoconference Care Management: 12-week nurse care management for medically complex Veterans with CI delivered via videoconferencing
  Care management via videoconference: 12-week nurse care management for medically complex Veterans with cognitive impairment delivered via videoconference
- Telephone Care Management: 12-week nurse care management for medically complex Veterans with CI delivered via telephone calls
  Care management via telephone calls: 12-week nurse care management for medically complex Veterans with cognitive impairment delivered via telephone calls
Period: Overall Study
Arm/Group | Videoconference Care Management | Telephone Care Management
Started | 40 (This number represents 20 dyads (1 Veteran and 1 caregiver in each dyad)) | 40 (This number represents 20 dyads (1 Veteran and 1 caregiver in each dyad))
Completed | 30 (This number represents 15 dyads (1 Veteran and 1 caregiver in each dyad)) | 32 (This number represents 16 dyads (1 Veteran and 1 caregiver in each dyad))
Not Completed | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Videoconference Care Management | Telephone Care Management | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The overall number of baseline participants differs from the number of analyzed participants because this study involved dyads (couples/pairs). Number analyzed in video intervention group=20 dyads (20 Veterans + 20 caregivers = 40 participants). Phone intervention group=20 dyads(20 Veterans + 20 caregivers = 40 participants).
  years
    Veterans: number analyzed (Participants) | 20 | 20 | 40
    Veterans | 70.2 (3.8) | 74.6 (7.1) | 72.4 (6.1)
    Caregivers: number analyzed (Participants) | 20 | 20 | 40
    Caregivers | 60.6 (12.0) | 68.9 (7.7) | 64.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The overall number of baseline participants differs from the number of analyzed participants because this study involved dyads (couples/pairs). Number analyzed in video intervention group=20 dyads (20 Veterans + 20 caregivers = 40 participants). Phone intervention group=20 dyads(20 Veterans + 20 caregivers = 40 participants).
  Participants
    Veterans: number analyzed (Participants) | 20 | 20 | 40
    Veterans: Female | 0 | 0 | 0
    Veterans: Male | 20 | 20 | 40
    Caregivers: number analyzed (Participants) | 20 | 20 | 40
    Caregivers: Female | 19 | 19 | 38
    Caregivers: Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The overall number of baseline participants differs from the number of analyzed participants because this study involved dyads (couples/pairs). Number analyzed in video intervention group=20 dyads (20 Veterans + 20 caregivers = 40 participants). Phone intervention group=20 dyads(20 Veterans + 20 caregivers = 40 participants).
  Participants
    Veterans: number analyzed (Participants) | 20 | 20 | 40
    Veterans: Hispanic or Latino | 0 | 0 | 0
    Veterans: Not Hispanic or Latino | 20 | 20 | 40
    Veterans: Unknown or Not Reported | 0 | 0 | 0
    Caregivers: number analyzed (Participants) | 20 | 20 | 40
    Caregivers: Hispanic or Latino | 0 | 0 | 0
    Caregivers: Not Hispanic or Latino | 20 | 20 | 40
    Caregivers: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The overall number of baseline participants differs from the number of analyzed participants because this study involved dyads (couples/pairs). Number analyzed in video intervention group=20 dyads (20 Veterans + 20 caregivers = 40 participants). Phone intervention group=20 dyads(20 Veterans + 20 caregivers = 40 participants).
  Participants
    Veterans: number analyzed (Participants) | 20 | 20 | 40
    Veterans: American Indian or Alaska Native | 0 | 0 | 0
    Veterans: Asian | 0 | 0 | 0
    Veterans: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Veterans: Black or African American | 8 | 7 | 15
    Veterans: White | 12 | 13 | 25
    Veterans: More than one race | 0 | 0 | 0
    Veterans: Unknown or Not Reported | 0 | 0 | 0
    Caregivers: number analyzed (Participants) | 20 | 20 | 40
    Caregivers: American Indian or Alaska Native | 0 | 0 | 0
    Caregivers: Asian | 0 | 0 | 0
    Caregivers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Caregivers: Black or African American | 8 | 3 | 11
    Caregivers: White | 12 | 17 | 29
    Caregivers: More than one race | 0 | 0 | 0
    Caregivers: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 40 | 80
Internet Use in Last Year [Count of Participants; unit: Participants] — Population: The overall number of baseline participants differs from the number of analyzed participants because this study involved dyads (couples/pairs). Number analyzed in video intervention group=20 dyads (20 Veterans + 20 caregivers = 40 participants). Phone intervention group=20 dyads(20 Veterans + 20 caregivers = 40 participants).
  Participants
    Veterans: number analyzed (Participants) | 20 | 20 | 40
    Veterans | 15 | 13 | 28
    Caregivers: number analyzed (Participants) | 20 | 20 | 40
    Caregivers | 19 | 13 | 32
Comfortable with Using the Internet [Count of Participants; unit: Participants] — Population: The overall number of baseline participants differs from the number of analyzed participants because this study involved dyads (couples/pairs). Number analyzed in video intervention group=20 dyads (20 Veterans + 20 caregivers = 40 participants). Phone intervention group=20 dyads(20 Veterans + 20 caregivers = 40 participants).
  Participants
    Veterans: number analyzed (Participants) | 20 | 20 | 40
    Veterans | 7 | 8 | 15
    Caregivers: number analyzed (Participants) | 20 | 20 | 40
    Caregivers | 16 | 11 | 27
Has Accessed Internet with Tablet Computer [Count of Participants; unit: Participants] — Population: The overall number of baseline participants differs from the number of analyzed participants because this study involved dyads (couples/pairs). Number analyzed in video intervention group=20 dyads (20 Veterans + 20 caregivers = 40 participants). Phone intervention group=20 dyads(20 Veterans + 20 caregivers = 40 participants).
  Participants
    Veterans: number analyzed (Participants) | 20 | 20 | 40
    Veterans | 4 | 2 | 6
    Caregivers: number analyzed (Participants) | 20 | 20 | 40
    Caregivers | 12 | 4 | 16
Previously Used Videochat [Count of Participants; unit: Participants] — Population: The overall number of baseline participants differs from the number of analyzed participants because this study involved dyads (couples/pairs). Number analyzed in video intervention group=20 dyads (20 Veterans + 20 caregivers = 40 participants). Phone intervention group=20 dyads(20 Veterans + 20 caregivers = 40 participants).
  Participants
    Veterans: number analyzed (Participants) | 20 | 20 | 40
    Veterans | 5 | 6 | 11
    Caregivers: number analyzed (Participants) | 20 | 20 | 40
    Caregivers | 13 | 10 | 23
Likely to see healthcare provider using videochat [Count of Participants; unit: Participants] — Population: The overall number of baseline participants differs from the number of analyzed participants because this study involved dyads (couples/pairs). Number analyzed in video intervention group=20 dyads (20 Veterans + 20 caregivers = 40 participants). Phone intervention group=20 dyads(20 Veterans + 20 caregivers = 40 participants).
  Participants
    Veterans: number analyzed (Participants) | 20 | 20 | 40
    Veterans | 11 | 8 | 19
    Caregivers: number analyzed (Participants) | 20 | 20 | 40
    Caregivers | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting That They Would Be Likely to See a Healthcare Provider Using Videochat
Description: Acceptability will be assessed using the measure of likelihood of seeing a healthcare provider using videochat.
Time Frame: 14 weeks
Population: These numbers represent the Veterans in the sample (Care Partners not analyzed)
Measure: Count of Participants; unit: Participants
Arm/Group | Videoconference Care Management | Telephone Care Management
Number analyzed (Participants) | 15 | 16
Participants | 6 | 5

2. Primary Outcome: Number of Scheduled Intervention Phone or Video Calls Completed by Participants
Description: Feasibility will be assessed by examining rates of adherence to intervention phone/video calls.
Time Frame: 14 weeks
Population: These number represent the Veterans in the sample (Care Partners not analyzed)
Measure: Count of Units; unit: calls
Units Other Than Participants: calls
Arm/Group | Videoconference Care Management | Telephone Care Management
Number analyzed (Participants) | 15 | 16
Number analyzed (calls) | 60 | 60
calls | 46 | 53

3. Primary Outcome: Usability of Video-Enhanced Care Management for Medically Complex Veterans With CI
Description: Usability of the video-enhanced care management program will be examined using the System Usability Scale (SUS; range 0 - 100; higher scores are better).
Time Frame: 14 weeks
Population: The System Usability Scale was administered only to the videoconference care management Veteran participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Videoconference Care Management | Telephone Care Management
Number analyzed (Participants) | 15 | 0
score on a scale | 59.3 (18.6) |

4. Other Pre Specified Outcome: Number of Participants With Hospitalizations or Emergency Department Visits
Description: Descriptive analysis of emergency department visits and hospitalizations in the two study arms
Time Frame: 14 weeks
Population: Utilization data was collected for Veteran participants only.
Measure: Number; unit: participants
Arm/Group | Videoconference Care Management | Telephone Care Management
Number analyzed (Participants) | 20 | 20
participants
  Hospitalizations | 2 | 1
  ED Visits | 4 | 1

5. Other Pre Specified Outcome: Physical Activity
Description: Descriptive analysis of physical activity as measured by the Physical Activity Scale for the Elderly (PASE; range 0 - 360; higher scores are better)
Time Frame: 14 weeks
Population: The PASE was administered to the Veteran participants only.
Measure: Mean (Standard Deviation); unit: weighted sum
Arm/Group | Videoconference Care Management | Telephone Care Management
Number analyzed (Participants) | 15 | 15
weighted sum | 75.1 (65.1) | 108.9 (73.8)

6. Other Pre Specified Outcome: Quality of Life Outcome
Description: Descriptive analysis of health-related quality of life as measured by 3 subscales of the Patient Reported Outcomes Measurement Information System (PROMIS-29; range 4 - 20 for each; lower scores are better)
Time Frame: 14 weeks
Population: The PROMIS subscales were administered to the Veteran participants only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Videoconference Care Management | Telephone Care Management
Number analyzed (Participants) | 15 | 15
score on a scale
  PROMIS-29 (Pain Interference) | 11.5 (5.7) | 10.9 (4.8)
  PROMIS-29 (Physical Function) | 12.3 (4.2) | 11.4 (5.5)
  PROMIS-29 (Social Roles) | 10.8 (3.8) | 11.5 (4.9)

7. Other Pre Specified Outcome: Depression
Description: Descriptive analysis of depression as measured by Patient Health Questionnaire-Depression (PHQ-9; range 0 - 27; lower scores are better)
Time Frame: 14 weeks
Population: The PHQ-9 was administered to the Veteran participants only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Videoconference Care Management | Telephone Care Management
Number analyzed (Participants) | 15 | 16
score on a scale | 6.4 (5.8) | 4.6 (3.7)

8. Other Pre Specified Outcome: Social Support
Description: Descriptive analysis of social support as measured by modified Medical Outcomes Study Social Support Survey (mMOS-SS; range 0 - 100; higher scores are better)
Time Frame: 14 weeks
Population: The mMOS-SS was administered to the Veteran participants only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Videoconference Care Management | Telephone Care Management
Number analyzed (Participants) | 15 | 15
score on a scale | 70.2 (26.0) | 72.7 (26.0)

9. Other Pre Specified Outcome: Anxiety
Description: Descriptive analysis of anxiety as measured by the Generalized Anxiety Disorder Scale (GAD-7; range 0 - 21; lower scores are better)
Time Frame: 14 weeks
Population: The GAD-7 was administered to the Veteran participants only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Videoconference Care Management | Telephone Care Management
Number analyzed (Participants) | 15 | 16
score on a scale | 4.2 (3.5) | 4.3 (3.8)

ADVERSE EVENTS:
Time Frame: 14 weeks
Groups:
- Videoconference Care Management - Veterans: 12-week nurse care management for medically complex Veterans with CI delivered via videoconferencing
  Care management via videoconference: 12-week nurse care management for medically complex Veterans with CI delivered via videoconference
- Telephone Care Management - Veterans: 12-week nurse care management for medically complex Veterans with CI delivered via telephone calls
  Care management via telephone calls: 12-week nurse care management for medically complex Veterans with CI delivered via telephone calls
- Videoconference Care Management - Care Partners: 12-week nurse care management for medically complex Veterans with CI and their care partners delivered via videoconferencing
  Care management via videoconference: 12-week nurse care management for medically complex Veterans with CI and their care partners delivered via videoconference
- Telephone Care Management - Care Partners: 12-week nurse care management for medically complex Veterans with CI and their care partners delivered via telephone calls
  Care management via telephone calls: 12-week nurse care management for medically complex Veterans with CI and their care partners delivered via telephone calls
Arm/Group | Videoconference Care Management - Veterans | Telephone Care Management - Veterans | Videoconference Care Management - Care Partners | Telephone Care Management - Care Partners
All-Cause Mortality (participants affected / at risk) | 1/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 4/20 | 3/20 | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Videoconference Care Management - Veterans (N=20) | Telephone Care Management - Veterans (N=20) | Videoconference Care Management - Care Partners (N=20) | Telephone Care Management - Care Partners (N=20)
Hospitalization (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Adverse events are reported as monitored/assessed
Hospitalization (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Adverse events are reported as monitored/assessed
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Videoconference Care Management - Veterans (N=20) | Telephone Care Management - Veterans (N=20) | Videoconference Care Management - Care Partners (N=20) | Telephone Care Management - Care Partners (N=20)
ED Visit (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) — Adverse events are reported as monitored/assessed
ED Visit (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Adverse events are reported as monitored/assessed
ED Visit (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Adverse events are reported as monitored/assessed
ED Visit (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Adverse events are reported as monitored/assessed
ED Visit (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Adverse events are reported as monitored/assessed

LIMITATIONS AND CAVEATS:
Perceived value associated with each delivery method was removed as an outcome on 2/13/19 because data are being analyzed as qualitative data; there are no quant data to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/87/NCT02962687/Prot_SAP_000.pdf